CLINICAL TRIAL: NCT03077568
Title: Evaluation of a Web Application That Supports Behavior Change in Work Related Stress - a Randomized Controlled Trial
Brief Title: Evaluation of a Web Application That Supports Behavior Change in Work Related Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/0646
Record Dates: First submitted 2016-12-07; First posted 2017-03-13 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Psychologic Stress; Occupation-Related Stress Disorder; Health Behavior
Keywords: internet; web-based; behavior change; stress-management
MeSH Terms: conditions — Stress, Psychological; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- My Stress Control (Experimental): This group gets access to the web-based program for stress-management. They will, by their own, go through the automated program. Measurements are conducted before, after as well as 3 months after the intervention.
  Interventions: Behavioral: My Stress Control
- Wait-list group (No Intervention): The wait-list grop will complete the same measures as the intervention group completes before and after the intervention with similar time spread. The wait-list group will then get access to the web-based program.

INTERVENTIONS:
Behavioral: My Stress Control — The web-based program is designed to educate the users in how stress can affect their health, provide tools to handle stress and also educate the users in a problem-solving method to prevent and manage stress-related problems in the future.
  The program is tailored for each user. The stress-management techniques included are: assertiveness training, change negative thinking, pleasant activity scheduling, relaxation, time-management, stimulus control and sleep restriction to improve sleep and physical activity.
  Central techniques to support behaivor change in My Stress Controll are encourage intention formulation, specific goal-setting, feedback on performance and reevaluation of goals.
  Arms: My Stress Control

SUMMARY:
A randomized controlled trial is needed to strengthen the evidence in the area of web-based self-management programs for stress-reduction.

Aim The aim for the study is to compare the effects of the web-application that supports behavior change in stress-management to a waiting list group in persons with perceived stress.

Method This study will have the design of a randomized controlled trial (RCT). The CONSORT guidelines will be used for reporting the study.

Sample: Different sectors in the region will be included. Three different high-schools in Västerås City, social services authority in Västerås municipality, a large private company in the region, three different clinics within the county council and the municipality of Köping have signed the attestation of participation.

Intervention: The intervention is the program for web-based stress self-management My Stress Control.

Procedure: After informed consent the participants will, during approximately 2-4 months by their own go through the web-based program for stress self-management. The waiting-list group will also get access to My Stress Control after post-measurements.

Data-analysis: Descriptive statistics will be used for demographic data. Missing data will be replaced as recommended for the different measurements included, commonly by using the mean for responded items within the sub scale. Inferential analyses will be conducted by using multivariate statistical analysis.

Drop-out analysis will be conducted by comparing pre-interventions measures for those who completed the program with those who did not.

DETAILED DESCRIPTION:
A randomized controlled trial is needed to strengthen the evidence in the area of web-based self-management programs for stress-reduction. The program to be evaluated is named My Stress Control, and is designed to educate the users in how stress can affect their health, provide tools to handle stress and also educate the users in a problem-solving method to prevent and manage stress-related problems in the future. My Stress Control is a self-administered and fully automated web-application.

Aim The aim for the study is to compare the effect of the web-application that supports behavior change in stress-management to a waiting list group in persons with perceived stress.

Method This study will have the design of a randomized controlled trial (RCT). The CONSORT guidelines will be used for reporting the study.

Sample: Different sectors in the region will be included. Three different high-schools in Västerås City, social services authority in Västerås municipality, a large private company in the region, three different clinics within the county council and the municipality of Köping have signed the attestation of participation.

Power: Power has been calculated by using a study comparing acceptance and commitment therapy with a wait-list group with the primary outcome stress, measured with PSS-14 (Cohen, Kamark, & Mermelstein, 1983). More specifically the power was calculated by using the scores of a group who reported lower stress-levels than 25 on PSS-14 (Brinkborg, Michaneck, Hessel, & Berglund, 2011). The calculation has been adjusted for both between-group comparison as well as for within-group comparison. An estimated effect size of .40 with power equal to .80 and a significance level of 0.05, gives an estimated population size of 98 individuals in each group. With an estimated dropout rate of 20% the population needed in each group is 118 persons.

Randomization: Since the included worksites are different to its kind, and to number of employees, randomization will be done by quotation with a 6-person block randomization. The block randomization will make the sample percentage similar to the included worksites.

Intervention: The intervention is the program for web-based stress self-management My Stress Control. My Stress Control starts with screening for stress levels according to Perceived Stress Scale (PSS) (Cohen et al., 1983), with a cut of score of 17 (Brinkborg et al., 2011) for accessing the program. To avoid to include users with more extended problems with anxiety and depression, a screening is done with Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983). Users scoring 11 or higher on either of the two subscales are recommended to seek support from traditional healthcare.

The security of the web-application is high and all information is encrypted. IP addresses who tries to log in without access are banned after a certain number of trials. The more secure https is used instead of the less secure http. All requests towards the server will be logged and all stored data have backup being done continuously.

Considering the theoretical framework of the self-management program there are several useful health psychological theories. Regarding behavior change in stress context three theories arise as more important; The Transactional Theory of Stress and Coping (TTC) (Lazarus & Folkman, 1984), Social Cognitive Theory (SCT) (Bandura, 1989), The Transtheoretical Model (TTM) and the Theory of Stages of Change (SoC) (Evers et al., 2006), and the Theory of Reasoned Action and the Theory of Planned Behavior(Madden, Ellen, & Ajzen, 1992). The theories play a crucial role in tailoring and assessing stress. Studies show that web-based programs using these theories are more successful than other web-based programs for behavior change (Webb, Joseph, Yardley, & Michie, 2010).

The program is sensitive to how the user formulates a guided functional behavior analysis that also tailors the program by recommending possible preferable stress-management techniques for each user. These stress-management techniques are specific behavior change techniques to support the user in situations where they experience stress or to prevent and handle consequences of stress. The user has the opportunity to take part of all stress-management techniques included.

The stress-management techniques included are: assertiveness training (Imamura et al., 2014), cognitive restructuring (Welbourne, Eggerth, Hartley, Andrew, & Sanches, 2007), pleasant activity scheduling (Mazzucchelli, Kane, & Rees, 2010), relaxation (Ponce et al., 2008), time-management (Häfner & Stock, 2010), stimulus control and sleep restriction to improve sleep (Thiart, Lehr, Ebert, Berking, & Riper, 2015) and physical activity (Lindegård, Jonsdottir, Börjesson, Lindwall, & Gerber, 2015). All techniques have shown to be effective in stress-management both in traditional face-to-face therapy and delivered in applications or on the web. Few programs have combined several techniques, and most programs use only one technique. No program combining all techniques included in My Stress Control has been found.

The most commonly used behavior modification techniques found in a meta-analysis of changing health behaviors via the Internet were to provide information about the consequences of the behavior, self-monitoring of behavior and identification of barriers and facilitators for behavior(Evers, Prochaska, Driskell, Cummins, & Velicer, 2003). In another study it is also stated that treatment that includes self-monitoring of the behavior and at least one of the following five behavioral change methods has been shown more effective than behavior modification treatment without these techniques; encourage intention formulation, specific goal-setting, feedback on performance and reevaluation of goals (Michie, Abraham, Whittington, McAteer, & Gupta, 2009). These techniques are central in the stress-management program. These behavior modification techniques are more general techniques for behavior change than the specific behavior change techniques for stress-management, and are used in several parts of My Stress Control. They are for example used to support the user to handle the specific techniques for stress management mentioned above. For example: Goal setting and self-monitoring is used as assignments in all the stress-management techniques in My Stress Control.

Thus, by using the web-based, self-management program My Stress Control, the individuals are supposed to receive support to develop skills to better cope with their work related stress.

Procedure: After informed consent the participants will, during approximately 2-4 months by their own go through the web-based program for stress self-management. The waiting-list group will also get access to My Stress Control after post-measurements. Reminders to send in the questionnaires will be sent out two weeks for the questionnaires answered before the intervention and two and four weeks after estimated time for the questionnaires answered during and after the intervention.

Data-analysis: Descriptive statistics will be used for demographic data. Missing data will be replaced as recommended for the different measurements included, commonly by using the mean for responded items within the sub scale. Inferential analyses will be conducted by using multivariate statistical analysis.

Drop-out analysis will be conducted by comparing pre-interventions measures for those who completed the program with those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Score 17 or more on Perceived Stress Scale -14
* Able to read and speak Swedish
* Employed
* Consent to take part in the study

Exclusion Criteria:

* Scoring 11 or more on either of sub scales of Hospital Anxiety and Depression Scale
* Currently on sick leave caused by stress, anxiety or depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in perceive stress measured with Perceived Stress Scale -14 | Before intervention, at intervention completion an average of 12 weeks, and for a 3 and 6 month follow up after completed intervention
  Wait-list group will conduct the same measures for their corresponding "pre" and "post" measures for an estimated timeframe of 2 months.

SECONDARY OUTCOMES:
Motivation for Change Questionnaire | Before intervention.
  Wait-list will complete this measure for their corresponding "pre"-measure
Change in self-efficacy believes for coping measured with Coping Self-Efficacy Scale | Before intervention, at intervention completion an average of 12 weeks, and for a 3 and 6 month follow up after completed intervention
  Wait-list group will conduct the same measures for their corresponding "pre" and "post" measures for an estimated timeframe of 2 months.
Change in perception of psychosocial factors at work measured with QPS Nordic-34+ for psychosocial factors at work | Before intervention, at intervention completion an average of 12 weeks, and for a 3 and 6 month follow up after completed intervention
  As Coping Self-Efficacy Scale
Change in work engagement measured with Utrecht work engagement Scale | Before intervention, at intervention completion an average of 12 weeks, and for a 3 and 6 month follow up after completed intervention
  As Coping Self-Efficacy Scale
Change in coping behaviors measured with Brief COPE Questionnaire | Before intervention, at intervention completion an average of 12 weeks, and for a 3 and 6 month follow up after completed intervention
  As Coping Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Anne Söderlund, PhD, Principal Investigator — Mälardalen University, Sweden
Locations (1):
- School of Health, Care and Social Welfare; Mälardalen University, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Bandura A. Human agency in social cognitive theory. Am Psychol. 1989 Sep;44(9):1175-84. doi: 10.1037/0003-066x.44.9.1175. PMID 2782727
- [Background] Brinkborg H, Michanek J, Hesser H, Berglund G. Acceptance and commitment therapy for the treatment of stress among social workers: a randomized controlled trial. Behav Res Ther. 2011 Jun;49(6-7):389-98. doi: 10.1016/j.brat.2011.03.009. Epub 2011 Apr 5. PMID 21513917
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Evers KE, Prochaska JM, Prochaska JO, Driskell MM, Cummins CO, Velicer WF. Strengths and weaknesses of health behavior change programs on the internet. J Health Psychol. 2003 Jan;8(1):63-70. doi: 10.1177/1359105303008001435. PMID 22113901
- [Background] Evers KE, Prochaska JO, Johnson JL, Mauriello LM, Padula JA, Prochaska JM. A randomized clinical trial of a population- and transtheoretical model-based stress-management intervention. Health Psychol. 2006 Jul;25(4):521-9. doi: 10.1037/0278-6133.25.4.521. PMID 16846327
- [Background] Hafner A, Stock A. Time management training and perceived control of time at work. J Psychol. 2010 Sep-Oct;144(5):429-47. doi: 10.1080/00223980.2010.496647. PMID 20806849
- [Background] Imamura K, Kawakami N, Furukawa TA, Matsuyama Y, Shimazu A, Umanodan R, Kawakami S, Kasai K. Effects of an Internet-based cognitive behavioral therapy (iCBT) program in Manga format on improving subthreshold depressive symptoms among healthy workers: a randomized controlled trial. PLoS One. 2014 May 20;9(5):e97167. doi: 10.1371/journal.pone.0097167. eCollection 2014. PMID 24844530
- [Background] Lazarus, R. S., & Folkman, S. (1984). Stress, appraisal and coping. New York, NY, US: Springer.
- [Background] Lindegard A, Jonsdottir IH, Borjesson M, Lindwall M, Gerber M. Changes in mental health in compliers and non-compliers with physical activity recommendations in patients with stress-related exhaustion. BMC Psychiatry. 2015 Nov 4;15:272. doi: 10.1186/s12888-015-0642-3. PMID 26530329
- [Background] Madden, T. J., Ellen, P. S., & Ajzen, I. (1992). A Comparison of the Theory of Planned Behavior and the Theory of Reasoned Action. Personality and Social Psychology Bulletin, 18(1), 3-9.
- [Background] Mazzucchelli TG, Kane RT, Rees CS. Behavioral activation interventions for well-being: A meta-analysis. J Posit Psychol. 2010 Mar;5(2):105-121. doi: 10.1080/17439760903569154. Epub 2010 May 7. PMID 20539837
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Ponce, A. N., Lorber, W., Paul, J. J., Esterlis, I., Barzvi, A., Allen, G. J., & Pescatello, L. S. (2008). Comparisons of Varying Dosages of Relaxation in a Corporate Setting: Effects on Stress Reduction. International Journal of Stress Management, 15(4), 396-407.
- [Background] Thiart H, Lehr D, Ebert DD, Berking M, Riper H. Log in and breathe out: internet-based recovery training for sleepless employees with work-related strain - results of a randomized controlled trial. Scand J Work Environ Health. 2015 Mar;41(2):164-74. doi: 10.5271/sjweh.3478. Epub 2015 Jan 15. PMID 25590336
- [Background] Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. J Med Internet Res. 2010 Feb 17;12(1):e4. doi: 10.2196/jmir.1376. PMID 20164043
- [Background] Welbourne, J. L., Eggerth, D., Hartley, T. A., Andrew, M. E., & Sanches, F. (2007). Coping strategies in the workplace: Relationships with attributional style and job satisfaction. . Journal of Vocational Behavior, 70(2), 312-325. doi:10.1016/j.jvb.2006.10.006
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Eklund C, Soderlund A, Elfstrom ML. Evaluation of a Web-Based Stress Management Program for Persons Experiencing Work-Related Stress in Sweden (My Stress Control): Randomized Controlled Trial. JMIR Ment Health. 2021 Dec 9;8(12):e17314. doi: 10.2196/17314. PMID 34889772